CLINICAL TRIAL: NCT06595329
Title: Comparison Between Epidural Analgesia and Intrathecal Opioid Analgesia for Pain Management in Open Nephrectomy: Prospective Randomized Controlled Trial
Brief Title: Comparison Between Epidural Analgesia and Intrathecal Opioid Analgesia for Pain Management in Open Nephrectomy
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital of Split (Other)
Responsible Party: Principal Investigator, Lenko Saric, Assistant professor, University Hospital of Split
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2181-147/01/06/LJ.Z.-23-04
Record Dates: First submitted 2024-08-27; First posted 2024-09-19 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Pain; Renal Cancer; Surgical Procedure, Unspecified
Keywords: Pain management; open nephrectomy; renal cell carcinoma
MeSH Terms: conditions — Pain; Kidney Neoplasms; Agnosia; Carcinoma, Renal Cell | interventions — Analgesia, Epidural

STUDY DESIGN:
Intervention Model Description: Prospective, single-center, randomized controlled trial. The study will take place in the University Hospital of Split, Departments of Anesthesiology, Reanimatology and Intensive Care Medicine, and the Department of Urology.
  Patients undergoing open radical or partial nephrectomy for renal cancer will be randomized to one of the two groups: Epidural analgesia (Control) or intrathecal opioid (Intervention) group. Physiologic functions (blood pressure, heart rate, peripheral oxygen saturation) will be monitored during and after the surgery. Postoperatively, pain scores at rest as well as during movement will be recorded. A total dose of intraoperative opioids, time to first rescue analgesic, and total dose of rescue analgesics as well as adverse effects during the first 72 hours postoperatively will be recorded. These parameters will be compared between the two groups.
Who Masked: Outcomes Assessor
Masking Description: Participants will be randomly divided into two groups in a 1:1 ratio. Randomization will be performed using a computer program. A research coordinator will be designated to distribute and preserve randomization results. A person designated for data analysis will be blinded for intervention performed in each group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Epidural analgesia (Active Comparator): An epidural catheter will be placed before induction to the anesthesia. A local anesthetic Levobupivacaine 0.25% (Levobupivakain Kabi ®, Fresenius Kabi Norge AS, Svinesundsveien, Norway, 5 mg/ml) will be administered as a bolus dose during the surgery and continuously (0.125% levobupivacaine) during the first 24 hours postoperatively. After the intervention, patients will undergo general anesthesia.
  Interventions: Procedure: Epidural analgesia
- Intrathecal opioid analgesia (Other): Patients in the Intervention group will receive a single dose of 300 mcg of morphine (Morphine Kalceks ®, Kalceks, AS, Riga, Latvija, 10mg/ml) intrathecally before induction to general anesthesia.
  Interventions: Procedure: Intrathecal opioid analgesia

INTERVENTIONS:
Procedure: Epidural analgesia — After establishing standard non-invasive monitoring of vital functions (electrocardiogram, blood pressure, peripheral oxygen saturation) and securing intravenous access, the patient will be seated. After sterile field preparation, a local anesthetic (2% lidocaine) will be administered at the site of the planned puncture. The epidural space will be identified at the level of the tenth thoracic intervertebral space using the loss of resistance technique and an 18G Tuohy epidural needle. After placing the epidural catheter, 4 ml of local anesthetic Levobupivacaine 0.25% will be administered into the epidural space. After inducing general anesthesia, an additional 4 ml of Levobupivacaine 0.25% will be administered before the surgical incision. Subjects in the control group will receive an infusion of 0.125% Levobupivacaine for 24 hours after the procedure.
  Arms: Epidural analgesia
Procedure: Intrathecal opioid analgesia — After establishing standard non-invasive monitoring of vital functions (electrocardiogram, blood pressure, peripheral oxygen saturation) and securing intravenous access, the patient will be seated. After sterile field preparation, a local anesthetic (2% lidocaine) will be administered at the site of the planned intrathecal puncture. Subsequently, at the selected site, the dura will be punctured using a spinal needle (25G Quincke spinal needle), and 0.3 mg of morphine will be administered to the patient. Following the intervention, the patient will be induced into general anesthesia.
  Other Names: Intrathecal morphine analgesia
  Arms: Intrathecal opioid analgesia

SUMMARY:
Nephrectomy is a surgical procedure of choice for patients suffering from renal cell carcinoma (RCC). Even though the laparoscopic approach is considered to cause fewer complications and reduce hospital stay, open surgery is still often performed. Open nephrectomy causes significant acute postoperative pain, and it can also lead to the development of chronic postoperative pain. Pain management is important for the overall recovery of patients undergoing major surgery such as open nephrectomy and it is a part of the enhanced recovery after surgery (ERAS) program.

In this prospective randomized clinical study, we plan to compare two different approaches to pain management regarding the level of acute pain (first 72 hours), side effects, systemic analgesics consumption, and hospital stay.

Our hypothesis are that intrathecal opioid administration significantly reduces acute postoperative pain compared to epidural analgesia in patients undergoing open radical or partial nephrectomy. We also hypothesize that the intrathecal opioid administration is associated with a lower incidence of adverse effects compared to epidural analgesia and shorter ICU length of stay.

DETAILED DESCRIPTION:
This is a prospective, single-center, randomized controlled trial. The study will take place in the University Hospital of Split, Departments of Anesthesiology, Reanimatology and Intensive Care Medicine, and the Department of Urology.

Patients undergoing open radical or partial nephrectomy for renal cancer will be randomized to one of the two groups: Epidural analgesia (Control) or intrathecal opioid (Intervention) group. Physiologic functions (blood pressure, heart rate, peripheral oxygen saturation) will be monitored during and after the surgery. Postoperatively, pain scores at rest as well as during movement will be recorded. A total dose of intraoperative opioids, time to first rescue analgesic, and total dose of rescue analgesics as well as adverse effects during the first 72 hours postoperatively will be recorded. These parameters will be compared between the two groups.

Data sources:

Patient records (electronic and paper), direct measurements of patients' physiologic functions (perioperatively, during first 72 hours postoperatively), pain assessment at rest, and movement (Numerical rating scale (NRS)).

Ways of collection of data:

Direct measurements will be used for physiologic functions (change in heart rate and blood pressure). NRS questionnaire will be used to measure pain at rest and during movement in the first 72 hours. Patient records will be used for demographic data and to measure side effects of the received treatment and length of ICU and hospital stay.

Measurements will be conducted by anesthesiologists in the operating room, staff in the ICU during the period we are investigating (72 hours after the procedure) and researchers going through patients' records.

The population represented by the sample:

Patients scheduled for open radical or partial nephrectomy due to RCC.

Independent variables:

Demographic data (age, gender, weight), comorbidities, chronic medication, chronic pain medication, American Society of Anesthesiologists (ASA) score, duration of surgery, duration of anesthesia, baseline NRS score.

Intervention group:

Patients with RCC undergoing open nephrectomy randomized into a group receiving intrathecal morphine.

Control group:

Patients who will receive epidural analgesia will be treated as a control group given that epidural analgesia is the most favorable analgesic technique in accordance with ERAS protocol for major abdominal surgeries.

Tehnique of randomisation:

Participants will be randomly divided into two groups in a 1:1 ratio. Randomization will be performed using a computer program. A research coordinator will be designated to distribute and preserve randomization results.

Patients with RCC undergoing open nephrectomy will be asked to sign written informed consent before the enrolment should they choose to participate in this study. They will be instructed on how to self-assess pain severity via the numeric rating scale before surgery (NRS, an 11-point scale where 0 = no pain and 10 = most severe pain).

Treatment/intervention:

Patients undergoing open radical or partial nephrectomy will randomly receive either epidural analgesia or intrathecal morphine.

Patients in the Intervention group will receive a single dose of 300 mcg of morphine intrathecally before induction to general anesthesia. For patients in the control group, an epidural catheter will be placed before induction to the anesthesia. A local anesthetic (levobupivacaine 0.25%) will be administered as a bolus dose during the surgery and continuously (0.125% levobupivacaine) during the first 24 hours postoperatively. After the intervention, patients will undergo general anesthesia.

Changes in heart rate, blood pressure, and the total dose of opioids administered are going to be measured intraoperatively. After the procedure, patients are going to be admitted to the intensive care unit in the Urology department. In the first 72 hours we will be measuring pain at rest using the Numerical rating scale (NRS), pain during cough using NRS, time of the first rescue analgesia, total dose of additional analgesics during 72 hours postoperatively, and the incidence of adverse effects (hypotension, bradycardia, nausea, vomiting, pruritus, respiratory insufficiency). We will analyze the quality of recovery and time to gastrointestinal function recovery. Complications of intervention will also be noted: accidental dural puncture, post-dural puncture headache, failed block, unintentional intravascular injection of local anesthetic, and local anesthetic toxicity. Length of ICU and hospital stay will also be measured. Patients will be exposed to intervention before the surgery, epidural catheter will be extracted after 24 hours. The expected duration of the study is one/two year/s.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients over the age of 18, scheduled for an open radical or partial nephrectomy due to RCC.
* American Society of Anesthesiologists (ASA) physical status classification I-III.

Exclusion Criteria:

* Patients who refuse to participate in this study.
* Patients with BMI > 35 kg/m2 or < 15 kg/m2.
* Patients with renal dysfunction (eGFR <15 or requirement of renal replacement therapy), liver dysfunction (Child-Pugh class C), and heart failure (NYHA IV).
* Patients with ASA physical status classification ≥ IV.
* Patients with contraindication for the interventions planned for in this study (allergies to anesthetic drugs used in this study, coagulation disorders, and infection at the injection site).
* Patients with chronic opioid dependence.
* Patients unable to communicate preoperatively due to severe dementia, language barrier, or neuropsychiatric disorder.
* Patients for whom it is impossible to carry out the aforementioned interventions for technical reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
NRS score at 24 hours postoperatively | 24 hours
  The primary outcome is the difference in NRS score at 24 hours postoperatively at rest and movement.
  Numeric rating scale (NRS) will be used, ranging from 0-10, where 0 means no pain and 10 means most severe pain.

SECONDARY OUTCOMES:
Intraoperative opioid consumption | Intraoperatively.
  Intraoperative opioid consumption in milligrams.
Numeric rating scale (NRS) score at 1, 3, 6, 48 and 72 hours postoperatively | 72 hours.
  Numeric rating scale (an 11-point scale where 0 = no pain and 10 = most severe pain) score at rest and movement at 1, 3, 6, 48, and 72 hours postoperatively.
Time to first rescue analgesia postoperatively | In the first 72 hours postoperatively.
  Time to first rescue analgesia postoperatively in hours.
Total amount of rescue analgesia during 24 and 72 hours postoperatively | 72 hours.
  Total amount of rescue analgesia during 24 and 72 hours postoperatively in mg.
Incidence of adverse effects | 72 hours.
  Incidence of adverse effects (hypotension defined as MAP ili SBP < 60 ili 90 mmHg for longer than 30 min), nausea, vomiting, accidental dural puncture with the needle or the catheter, post-dural puncture headache (headache occurring within 5 days after a lumbar puncture, accompanied by neck stiffness and subjective changes in hearing), failed block (total absence of any neuraxial block or the development of a partial block that is of insufficient height, duration, or quality), unintentional intravascular injection of local anesthetic, local anesthetic toxicity and respiratory depression (respiratory rate ≤8 breaths/min).
Duration of procedure performance | During procedure execution (epidural catether placement, intrathecal administration of the drug).
  Duration of procedure performance from the administration of local anesthetic for skin puncture to the removal of epidural or spinal needle in minutes.
Gastrointestinal function recovery | Up to 72 hours post operatively.
  Gastrointestinal function recovery time (time to first bowel movement) in hours.
Hospital length of stay | Through study completion, an average of 1 year.
  Hospital length of stay in days.
ICU length of stay | Through study completion, an average of 1 year.
  ICU length of stay in days.

CONTACTS AND LOCATIONS:
Overall Officials: Svjetlana Došenović, MD Phd, Principal Investigator — UH Split
Locations (1):
- Univeristy Hospital of Split, Split, Croatia

IPD SHARING:
Plan to Share IPD: Undecided